CLINICAL TRIAL: NCT02553499
Title: A Phase 1 Trial of MK-1248 as Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors.
Brief Title: Study of MK-1248 With and Without Pembrolizumab (MK-3475) for Participants With Advanced Solid Tumors (MK-1248-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment prematurely discontinued due to program prioritization & not due to any safety concerns.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1248-001; MK-1248-001 (Other: Merck)
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Advanced Solid Tumor
Keywords: Solid tumor; PD1; PD-L1; PDL1
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-1248 (Experimental): Participants received escalating doses of MK-1248 at assigned dose (dose range: 0.12 mg to 170 mg MK-1248) via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to ~3 months).
  Interventions: Biological: MK-1248
- MK-1248 + Pembrolizumab (Experimental): Participants received escalating doses of MK-1248 at assigned dose (dose range: 0.12 mg to 60 mg MK-1248) via IV infusion on Day 1 of each 21-day cycle for a maximum of 4 cycles (up to ~3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~24 months).
  Interventions: Biological: MK-1248; Biological: pembrolizumab

INTERVENTIONS:
Biological: MK-1248 — IV infusion
Biological: pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: MK-1248 + Pembrolizumab

SUMMARY:
In this study, participants with advanced solid tumors were assigned to receive escalating doses of either MK-1248 alone or MK-1248 in combination with pembrolizumab (MK-3475). This study used the number of dose-limiting toxicities (DLTs) at each dose level to find and confirm the maximum tolerated dose (or maximum administered dose) for MK-1248 alone and in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed metastatic solid tumor for which there is no available therapy that may convey clinical benefit
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Adequate organ function
* Female participants of childbearing potential should be willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication
* Male participants should agree to use adequate contraception starting with the first dose of study therapy through 180 days after the last dose of study medication
* Can submit a baseline tumor sample

Exclusion Criteria:

* Has had chemotherapy, radiation, or biological cancer therapy within 4 weeks prior to the first dose of study medication, or not recovered from adverse events due to cancer therapeutics administered more than 4 weeks earlier
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study medication
* Previous treatment with another agent targeting the glucocorticoid-induced tumor necrosis factor receptor-related protein (GITR) receptor
* Previous treatment with an immunomodulatory therapy and was discontinued from that therapy due to an immune-related adverse event
* Expected to require any other form of antineoplastic therapy while on study
* On chronic systemic steroid therapy in excess of replacement doses, or on any other form of immunosuppressive medication
* History of a previous, additional malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 5 years with the exception of successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Severe hypersensitivity reaction to treatment with another monoclonal antibody
* Active autoimmune disease or a documented history of autoimmune disease with the exception of vitiligo or resolved childhood asthma/atopy, or endocrine deficiency following treatment with an immunomodulatory agent
* Active infection requiring therapy
* Active or a history of non-infectious pneumonitis
* Prior stem cell or bone marrow transplant
* Known history of human immunodeficiency virus (HIV), active chronic or acute hepatitis B or C
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol), at the time of signing informed consent
* Symptomatic ascites or pleural effusion
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study through 180 days after the last dose of study medication
* Major surgery within 16 weeks prior to screening
* Live vaccine within 30 days prior to first dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Geva R, Voskoboynik M, Dobrenkov K, Mayawala K, Gwo J, Wnek R, Chartash E, Long GV. First-in-human phase 1 study of MK-1248, an anti-glucocorticoid-induced tumor necrosis factor receptor agonist monoclonal antibody, as monotherapy or with pembrolizumab in patients with advanced solid tumors. Cancer. 2020 Nov 15;126(22):4926-4935. doi: 10.1002/cncr.33133. Epub 2020 Aug 18. PMID 32809217

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-1248 0.12 mg: Participants received MK-1248 0.12 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 0.6 mg: Participants received MK-1248 0.6 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 3 mg: Participants received MK-1248 3 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 10 mg: Participants received MK-1248 10 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 30 mg: Participants received MK-1248 30 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 60 mg: Participants received MK-1248 60 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 120 mg: Participants received MK-1248 120 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 170 mg: Participants received MK-1248 170 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- MK-1248 0.12 mg + Pembrolizumab: Participants received MK-1248 0.12 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 24 months).
- MK-1248 0.6 mg + Pembrolizumab: Participants received MK-1248 0.6 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 24 months).
- MK-1248 3 mg + Pembrolizumab: Participants received MK-1248 3 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 24 months).
- MK-1248 10 mg + Pembrolizumab: Participants received MK-1248 10 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 24 months).
- MK-1248 30 mg + Pembrolizumab: Participants received MK-1248 30 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 24 months).
- MK-1248 60 mg + Pembrolizumab: Participants received MK-1248 60 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months) PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 24 months).
Period: Overall Study
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Started | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-1248 0.12 mg: Participants received MK-1248 0.12 mg via IV infusion on Day 1 of each 21-day cycle for up to 4 cycles (up to approximately 3 months).
- Total: Total of all reporting groups
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (1.4) | 43.5 (3.5) | 58.5 (12.9) | 49.5 (17.7) | 63.7 (3.8) | 50.3 (14.0) | 58.3 (3.1) | 69.3 (6.0) | 54.0 (19.1) | 77.3 (8.7) | 57.7 (5.0) | 71.3 (8.6) | 51.7 (7.5) | 72.5 (7.8) | 60.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 15
  Male | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 3 | 3 | 1 | 2 | 2 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose-Limiting Toxicity (DLT)
Description: The occurrence of any of the following toxicities during Cycle 1 (21 days), if possibly, probably or definitely related to study treatment, was considered a DLT: 1. Grade 4 non-hematological toxicity 2. Grade 4 hematological toxicity lasting >7 days, except thrombocytopenia a. Grade 4 thrombocytopenia of any duration b. Grade 3 thrombocytopenia is a DLT if associated with bleeding 3. Any Grade 3 non-hematological toxicity, with the exceptions 4. Any Grade 3 or Grade 4 non-hematological laboratory abnormality, if medical intervention was required, or abnormality led to hospitalization, or abnormality persisted for >1 week 5. Febrile neutropenia Grade 3 or Grade 4 6. Any drug-related AE which caused participant to discontinue study treatment during Cycle 1 7. Grade 5 toxicity 8. Any treatment-related toxicity which caused a >2-week delay in initiation of Cycle 2.
Time Frame: Cycle 1 (Up to 21 days)
Population: The DLT analysis population consisted of all participants who received MK-1248 and were observed for safety for 21 days after the first dose of MK-1248 or experienced a DLT prior to 21 days after the first dose of MK-1248.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Concentration (Cmax) of MK-1248 in Serum
Description: Cmax is the maximum (peak) concentration of MK-1248 observed in blood serum. Blood samples were obtained at designated timepoints for the analysis of MK-1248 Cmax. Timepoints: Cycles 1-4 Day 1: Predose, post MK-1248 infusion end (~0.5 hours), 2 hours post MK-1248 infusion start (~2 hours); Cycles 1-4 Days 2, 3, 5, 8 & 15. Each cycle was 21 days. (Up to ~3 months)
Time Frame: At designated timepoints (Up to ~3 months)
Population: The analysis population consisted of all participants who received MK-1248 and had blood samples assessed for MK-1248 Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
pg/mL
  Cycle 1 | 45800 (82.5) | 378000 (63.9) | 853000 (19.9) | 3550000 (23.1) | 10200000 (39.0) | 13300000 (110.7) | 38600000 (32.8) | 59400000 (12.2) | 69500 (32.7) | 567000 (650.2) | 820000 (51.4) | 4360000 (21.0) | 8710000 (42.8) | 12900000 (44.8)
  Cycle 2: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 1
  Cycle 2 | 112000 (27.0) | 154000 (247.8) | 1260000 (69.1) | 186000 (1615.9) | 8590000 (64.1) | 6240000 (481.2) | 41500000 (40.0) | 6980000 (24178.9) | 41900 (28.5) | 141000 (13.5) | 981000 (17.7) | 1950000 (14.3) | 10400000 (43.4) | 16900000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 3: number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 3 | 2 | 3 | 3 | 2 | 1
  Cycle 3 | 17600 (312.1) | 52400 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 842000 (16.5) | 843000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 10200000 (65.9) | 21500000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 52600000 (46.9) | 67400000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 170000 (284.4) | 136000 (59.4) | 891000 (37.1) | 2270000 (39.8) | 12300000 (30.3) | 16100000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 4: number analyzed (Participants) | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 2 | 2 | 1
  Cycle 4 | 1000000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 5090 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 566000 (45.8) |  | 17100000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 12600000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 70700000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 66300000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 76300 (320.4) | 3460 (229.1) | 568000 (224.7) | 911000 (481.5) | 12200000 (45.2) | 12800000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant

3. Secondary Outcome: Trough Concentration (Ctrough) of MK-1248 in Serum
Description: Ctrough is the lowest concentration of MK-1248 in blood serum just before the next dose. Blood samples were obtained at designated timepoints for the analysis of MK-1248 Ctrough, except for during Cycle 1. No blood samples were collected for the analysis of Ctrough in Cycle 1. No samples were collected for the MK-1248 0.6 mg group in Cycles 3 or 4, for the MK-1248 10 mg group in Cycles 1-4, or for the MK-1248 60 mg + Pembrolizumab group in Cycle 4. Timepoints: Cycles 1-4 Day 1: Predose, post MK-1248 infusion end (~0.5 hours), 2 hours post MK-1248 infusion start (~2 hours); Cycles 1-4 Days 2, 3, 5, 8 & 15. Each cycle was 21 days. (Up to ~3 months)
Time Frame: At designated timepoints (Up to ~3 months)
Population: The analysis population consisted of all participants who received MK-1248 and had blood samples assessed for MK-1248 Ctrough. Ctrough data were not collected for the MK-1248 10 mg group
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
pg/mL
  Cycle 1: number analyzed (Participants) | 2 | 1 | 1 | 0 | 2 | 3 | 3 | 1 | 3 | 3 | 1 | 0 | 3 | 1
  Cycle 1 | 74.1 (186.2) | 427 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 14100 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 767000 (798.2) | 282000 (1824.0) | 1290000 (21562.3) | 4660000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 56.2 (142.3) | 98.1 (28.4) | 18400 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 345000 (2621.6) | 1830000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 2: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 3 | 1
  Cycle 2 | 106 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 23900 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 485000 (24904.1) | 112000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 9530000 (130.5) | 828000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 41.0 (95.6) |  |  |  | 2180000 (130.0) | 295000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 3: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1
  Cycle 3 | 102 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 14200 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 6840000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 123000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 25600000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 119000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 48.8 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  |  |  | 1670000 (290.5) | 15700 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Cycle 4 |  |  |  |  |  |  |  |  | 25.1 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  |  |  | 4830000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |

4. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to Infinity (AUC0-inf) of MK-1248 in Serum
Description: AUC0-infinity is the area under the serum concentration-time curve from time zero to infinity. It is a measure of the amount of MK-1248 in blood serum from pre-dose to infinite time. Blood samples were obtained at designated timepoints for the analysis of MK-1248 AUC0-inf. No blood samples were collected for the MK-1248 0.6 mg group in Cycle 4, for the MK-1248 10 mg group in Cycle or for the MK-1248 60 mg + Pembrolizumab group in Cycle 4. Timepoints: Cycles 1-4 Day 1: Predose, post MK-1248 infusion end (~0.5 hours), 2 hours post MK-1248 infusion start (~2 hours); Cycles 1-4 Days 2, 3, 5, 8 & 15. Each cycle was 21 days. (Up to ~3 months)
Time Frame: At designated timepoints (Up to ~3 months)
Population: The analysis population consisted of all participants who received MK-1248 and had blood samples assessed for MK-1248 AUC0-inf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*pg/mL
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Days*pg/mL
  Cycle 1: number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
  Cycle 1 | 99200 (123.5) | 1010000 (70.8) | 4390000 (24.9) | 25100000 (3.6) | 117000000 (57.5) | 175000000 (26.0) | 354000000 (73.5) | 596000000 (34.2) | 78000 (9.4) | 608000 (14.3) | 3260000 (78.8) | 28100000 (27.5) | 77900000 (89.3) | 128000000 (28.2)
  Cycle 2: number analyzed (Participants) | 2 | 2 | 2 | 0 | 2 | 2 | 2 | 1 | 3 | 3 | 3 | 0 | 3 | 1
  Cycle 2 | 120000 (40.8) | 77200 (5679.1) | 5600000 (24.1) |  | 84200000 (618.4) | 105000000 (304.5) | 604000000 (111.5) | 341000000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 80400 (70.4) | 273000 (33.3) | 3860000 (44.1) |  | 64900000 (285.6) | 77300000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 3: number analyzed (Participants) | 1 | 0 | 2 | 0 | 2 | 1 | 2 | 1 | 3 | 2 | 3 | 2 | 2 | 1
  Cycle 3 | 91700 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 1770000 (212.1) |  | 124000000 (783.4) | 50500000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 737000000 (172.7) | 218000000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 393000 (1325.8) | 94300 (76.7) | 1010000 (79.4) | 802000 (289.8) | 139000000 (125.9) | 31500000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant
  Cycle 4: number analyzed (Participants) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 3 | 1 | 2 | 1
  Cycle 4 |  |  | 864000 (439.4) |  | 460000000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 21200000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 1440000000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 250000000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 84300 (378.0) |  | 295000 (347.2) | 3040000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 112000000 (259.6) | 22100000 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant

5. Secondary Outcome: Maximum Concentration (Cmax) of Glucocorticoid-induced Tumor Necrosis Factor Receptor-related Protein (GITR) Receptor Target Engagement
Description: GITR protein is internalized upon binding by MK-1248. To evaluate GITR target engagement, a GITR receptor availability assay was developed to assess the availability of surface GITR following administration of MK-1248. GITR is detected on CD4+CD25+ and CD4+CD95+ T-cell sub-populations using flow cytometry and compared to pre-dose baseline. GITR target engagement is calculated as 100% - (%) GITR receptor availability. The Cmax of percent GITR target engagement on CD4+CD25+ T-cells is presented. Timepoints: Arm 1: Screening; Cycles 1-4 Day 1: Predose MK-1248, At end of MK-1248 infusion (0.5 hours), 2 hours after start of MK-1248 infusion (2 hours); Cycles 1-4 Days 2, 8 & 15. Arm 2: Screening; Cycles 1-4 Day 1: Predose pembrolizumab, At end of MK-1248 infusion (0.5 hours), 2 hours after start of MK-1248 infusion (2 hours): Cycles 1-4 Days 2, 3, 8 & Day 15: Cycles 5-6: Predose. Each cycle was 21 days.
Time Frame: At designated timepoints (Up to ~4.5 months)
Population: The analysis population consisted of all participants who received MK-1248 and had blood samples assessed for GITR receptor target engagement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent Target Engagement
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Number analyzed (Participants) | 2 | 1 | 2 | 0 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2
Percent Target Engagement | 32.1 (141.4) | 83.8 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 94.5 (7.8) |  | 84.5 (13.5) | 69.7 (29.6) | 96.8 (1.9) | 47.3 (58.0) | 71.6 (20.4) | 89.3 (6.2) | 89.9 (7.8) | 68.9 (41.5) | 80.8 (24.7) | 68.0 (46.3)

6. Secondary Outcome: Trough (Minimum) Concentration (Ctrough) of Glucocorticoid-induced Tumor Necrosis Factor Receptor-related Protein (GITR) Receptor Target Engagement
Description: GITR protein is internalized upon binding by MK-1248. To evaluate GITR target engagement, a GITR receptor availability assay was developed to assess the availability of surface GITR following administration of MK-1248. GITR is detected on CD4+CD25+ and CD4+CD95+ T-cell sub-populations using flow cytometry and compared to pre-dose baseline. GITR target engagement is calculated as 100% - (%) GITR receptor availability. The Ctrough of percent GITR target engagement on CD4+CD25+ T-cells is presented. Timepoints: Arm 1: Screening; Cycles 1-4 Day 1: Predose MK-1248, At end of MK-1248 infusion (0.5 hours), 2 hours after start of MK-1248 infusion (2 hours); Cycles 1-4 Days 2, 8 & 15. Arm 2: Screening; Cycles 1-4 Day 1: Predose pembrolizumab, At end of MK-1248 infusion (0.5 hours), 2 hours after start of MK-1248 infusion (2 hours): Cycles 1-4 Days 2, 3, 8 & Day 15: Cycles 5-6: Predose. Each cycle was 21 days.
Time Frame: At designated timepoints (Up to ~4.5 months)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent Target Engagement
Groups:
- MK-1248 170 mg: Participants received MK-1248 at selected monotherapy dose (170 mg) via IV infusion on Day 1 of each 21-day cycle for a maximum of 4 cycles (up to ~3 months).
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
Number analyzed (Participants) | 2 | 1 | 1 | 0 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 2
Percent Target Engagement | 3.2 (141.4) | 36.6 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 48.9 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant |  | 94.0 (2.1) | 83.7 (23.0) | 89.1 (5.4) | 57.3 (50.8) | 33.7 (4.0) | 6.2 (95.2) | 88.7 (3.6) | 5.9 (173.2) | 96.7 (NA) — NA=Geometric Coefficient of Variation could not be calculated with only 1 participant | 70.2 (2.6)

ADVERSE EVENTS:
Time Frame: Up to ~27 months
Description: Safety Population: All participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered an adverse event (AE) unless considered related to study treatment. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | MK-1248 0.12 mg | MK-1248 0.6 mg | MK-1248 3 mg | MK-1248 10 mg | MK-1248 30 mg | MK-1248 60 mg | MK-1248 120 mg | MK-1248 170 mg | MK-1248 0.12 mg + Pembrolizumab | MK-1248 0.6 mg + Pembrolizumab | MK-1248 3 mg + Pembrolizumab | MK-1248 10 mg + Pembrolizumab | MK-1248 30 mg + Pembrolizumab | MK-1248 60 mg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/2 | 2/2 | 0/2 | 3/3 | 2/3 | 1/3 | 3/3 | 2/3 | 0/3 | 1/3 | 2/3 | 1/3 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 0/2 | 0/2 | 0/3 | 1/3 | 2/3 | 1/3 | 1/3 | 2/3 | 0/3 | 2/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1248 0.12 mg (N=2) | MK-1248 0.6 mg (N=2) | MK-1248 3 mg (N=2) | MK-1248 10 mg (N=2) | MK-1248 30 mg (N=3) | MK-1248 60 mg (N=3) | MK-1248 120 mg (N=3) | MK-1248 170 mg (N=3) | MK-1248 0.12 mg + Pembrolizumab (N=3) | MK-1248 0.6 mg + Pembrolizumab (N=3) | MK-1248 3 mg + Pembrolizumab (N=3) | MK-1248 10 mg + Pembrolizumab (N=3) | MK-1248 30 mg + Pembrolizumab (N=3) | MK-1248 60 mg + Pembrolizumab (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1248 0.12 mg (N=2) | MK-1248 0.6 mg (N=2) | MK-1248 3 mg (N=2) | MK-1248 10 mg (N=2) | MK-1248 30 mg (N=3) | MK-1248 60 mg (N=3) | MK-1248 120 mg (N=3) | MK-1248 170 mg (N=3) | MK-1248 0.12 mg + Pembrolizumab (N=3) | MK-1248 0.6 mg + Pembrolizumab (N=3) | MK-1248 3 mg + Pembrolizumab (N=3) | MK-1248 10 mg + Pembrolizumab (N=3) | MK-1248 30 mg + Pembrolizumab (N=3) | MK-1248 60 mg + Pembrolizumab (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment into this study was prematurely discontinued due to program prioritization and not related to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT02553499/Prot_SAP_000.pdf